CLINICAL TRIAL: NCT01954342
Title: MomEE: Determinants of Gestational Weight Gain in Obese Pregnant Women
Brief Title: Determinants of Gestational Weight Gain in Obese Pregnant Women
Acronym: MomEE
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 13020; 1R01DK099175 (NIH)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Energy Intake; Energy Expenditure
Keywords: Pregnancy; Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Placenta, Cord Blood, fasting Urine, fasting Maternal plasma and serum (during pregnancy and postpartum).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant: Obese pregnant women

SUMMARY:
The purpose of this study is to measure energy intake and energy expenditure during and after pregnancy. The investigators hypothesize that obese pregnant women with weight gain above the Institute of Medicine (IOM) guidelines, 'High Gainers', will have increased energy intake but no evidence for changes in energy expenditure after adjustment for the weight gained when compared to women with appropriate gestational weight gain, 'Normal Gainers'. Additionally, the investigators will measure the babies born to the pregnant women enrolled in MomEE at one time point before 10 days of life.

ELIGIBILITY:
Inclusion Criteria:

* Are pregnant
* Have a body mass index (BMI) greater than or equal to 30kg/m2
* Are 18-40 years old
* Medically cleared for participation by primary care obstetrician
* Medically cleared for participant by Medical Investigator
* Willingness to allow the study access to information in the participant's medical record
* Willingness to be notified of incidental findings from study procedures

Exclusion Criteria:

Clinical

* Hypertension (i.e. systolic blood pressure (SBP) >160 mmHg & diastolic blood pressure (DBP) >110 mmHg)*
* Diagnosis of diabetes prior to pregnancy
* Hb A1c ≥6.5 %*
* Implanted metal objects that render MRI unsafe
* HIV or AIDS (self-reported)
* Severe anemia (hemoglobin <8g/dL and/or hematocrit <24%)** Psychological
* History or current psychotic disorder or diagnosis of a current major depressive episode or bipolar disorder
* Past history of anorexia or bulimia by medical history or patient report (binge eating disorder is not an exclusion) or current eating disorder
* Actively suicidal defined as a value ≥2 on the Beck Depression Index (BDI-II) question 9* Medications
* Current use of one or more of the following medications: metformin, systemic steroids, antipsychotic agents (e.g., Abilify, Haldol, Risperdal, Seroquel, Zyprexa), anti-seizure medications or mood stabilizers that would be expected to have a significant impact on body weight (e.g., Depakote, Lamictal, Lithium, Neurontin, Tegretol, Topamax, Keppra), medications for attention-deficit/hyperactivity disorder (ADHD) including amphetamines and methylphenidate
* Continued use of weight loss medication including over the counter (OTC) and dietary supplements for weight loss (e.g., Adipex, Suprenza, Tenuate, Xenical, Alli, conjugated linoleic acid, Hoodia, Green tea extract, Guar gum, HydroxyCut, Sensa, Corti-slim, Chromium, chitosan, Bitter orange) Other Exclusion Criteria
* Recent history of or currently smoking, drinking alcohol or abusing drugs (prescription or recreational)
* Plans to move out of the study area within the next 2 years or plans to be out of the study area for more than 4 weeks in the next 12 months
* Planned termination of pregnancy
* Unwillingness to avoid pregnancy for 12 months following delivery
* Claustrophobia
* Prior or planned (within 1 year of expected delivery) bariatric surgery
* Participant's unwillingness or inability to commit to a 1 year follow-up

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 75 obese, pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, PhD, Principal Investigator — Pennington Biomedical Research
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Lindsay KL, Most J, Buehler K, Kebbe M, Altazan AD, Redman LM. Maternal mindful eating as a target for improving metabolic outcomes in pregnant women with obesity. Front Biosci (Landmark Ed). 2021 Dec 30;26(12):1548-1558. doi: 10.52586/5048. PMID 34994169
- [Derived] Most J, Altazan AD, St Amant M, Beyl RA, Ravussin E, Redman LM. Increased Energy Intake After Pregnancy Determines Postpartum Weight Retention in Women With Obesity. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1601-11. doi: 10.1210/clinem/dgz330. PMID 31905403
- [Derived] Most J, Amant MS, Hsia DS, Altazan AD, Thomas DM, Gilmore LA, Vallo PM, Beyl RA, Ravussin E, Redman LM. Evidence-based recommendations for energy intake in pregnant women with obesity. J Clin Invest. 2019 Aug 1;129(11):4682-4690. doi: 10.1172/JCI130341. PMID 31369400
- [Derived] Most J, Redman LM. Energy expenditure predictions in postpartum women require adjustment for race. Am J Clin Nutr. 2019 Aug 1;110(2):522-524. doi: 10.1093/ajcn/nqz087. No abstract available. PMID 31367759
- [Derived] Most J, Vallo PM, Gilmore LA, St Amant M, Hsia DS, Altazan AD, Beyl RA, Ravussin E, Redman LM. Energy Expenditure in Pregnant Women with Obesity Does Not Support Energy Intake Recommendations. Obesity (Silver Spring). 2018 Jun;26(6):992-999. doi: 10.1002/oby.22194. PMID 29797559
- [Derived] Most J, Gilmore LA, Altazan AD, St Amant M, Beyl RA, Ravussin E, Redman LM. Propensity for adverse pregnancy outcomes in African-American women may be explained by low energy expenditure in early pregnancy. Am J Clin Nutr. 2018 Jun 1;107(6):957-964. doi: 10.1093/ajcn/nqy053. PMID 29767680
- [Derived] Most J, Vallo PM, Altazan AD, Gilmore LA, Sutton EF, Cain LE, Burton JH, Martin CK, Redman LM. Food Photography Is Not an Accurate Measure of Energy Intake in Obese, Pregnant Women. J Nutr. 2018 Apr 1;148(4):658-663. doi: 10.1093/jn/nxy009. PMID 29659958
- [Derived] Sutton EF, Cain LE, Vallo PM, Redman LM. Strategies for Successful Recruitment of Pregnant Patients Into Clinical Trials. Obstet Gynecol. 2017 Mar;129(3):554-559. doi: 10.1097/AOG.0000000000001900. PMID 28178062
- See also: Reproductive Endocrinology & Women's Health Laboratory- Our Research — http://labs.pbrc.edu/womenshealth/research.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Women With Excess Gestational Weight Gain: Pregnant women with weight gain above the Institutes of Medicine gestational weight gain guidelines
- Pregnant Women With Recommended Gestational Weight Gain: Pregnant women with weight gain within the Institutes of Medicine gestational weight gain guidelines
- Pregnant Women With Inadequate Gestational Weight Gain: Pregnant women with weight gain below the Institutes of Medicine gestational weight gain guidelines
- Pregnant Women Not Included in Analysis: Pregnant women who enrolled in the study but were not included in data analysis for various reasons.
Period: Overall Study
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Started | 36 | 8 | 10 | 18
Completed | 36 | 8 | 10 | 0
Not Completed | 0 | 0 | 0 | 18
Not completed — Missing data from 13-16week study visit | 0 | 0 | 0 | 1
Not completed — Miscarriage | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5
Not completed — Preterm delivery | 0 | 0 | 0 | 3
Not completed — Pre-eclampsia | 0 | 0 | 0 | 4
Not completed — Unreliable Data | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis | Total
Number analyzed (Participants) | 36 | 8 | 10 | 18 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (4.8) | 25 (4.8) | 29.2 (4.1) | 28.2 (6.1) | 27.7 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 8 | 10 | 18 | 72
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 4 | 6 | 12 | 34
  White | 22 | 3 | 3 | 4 | 32
  More than one race | 1 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Parity [Count of Participants; unit: Participants]
  0 viable pregnancies | 16 | 4 | 3 | 11 | 34
  1 viable pregnancies | 14 | 2 | 3 | 3 | 22
  2 viable pregnancies | 4 | 1 | 3 | 2 | 10
  ≥3 viable pregnancies | 2 | 1 | 1 | 2 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.8 (3.0) | 34.6 (4.5) | 40.6 (7.9) | 41.0 (6.3) | 37.1 (5.7)
Highest Education [Count of Participants; unit: Participants]
  Less than high school | 0 | 0 | 0 | 1 | 1
  High school | 6 | 1 | 1 | 1 | 9
  1-3 years college | 11 | 3 | 4 | 13 | 31
  College degree | 10 | 4 | 2 | 2 | 18
  Postgraduate work | 9 | 0 | 3 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Energy Intake
Description: Energy intake is determined using the energy intake-balance method. Energy intake was calculated as the sum of energy expenditure by doubly labeled water and energy deposition of fat and fat-free tissues by 3 compartment model using plethysmography and isotope dilution.
Time Frame: Approximately 6 months (from 13-16 weeks gestation to 35-37 weeks gestation)
Population: Analysis could not be completed for the Arm (Pregnant Women Not Included in Analysis). Reasons include the following: missing necessary data from either the 13-16 weeks gestation or 35-37 weeks gestation visit, pre-eclampsia, or unreliable data.
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 36 | 8 | 10 | 0
kilocalories per day | 2908 (384) | 2698 (280) | 2581 (417) |

2. Secondary Outcome: Physical Activity
Description: Physical activity is determined using daily mean amplitude deviation in milligrams by wrist worn accelerometer over a period of approximately 7 days within early pregnancy (13-16 weeks gestation). Mean amplitude deviation describes the mean distance of data points from the mean, and higher values denote higher levels of physical activity.
Time Frame: Approximately 7 days within 13-16 weeks gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 36 | 8 | 10 | 0
milligrams | 53.8 (10.2) | 56.4 (6.5) | 46.6 (9.8) |

3. Secondary Outcome: Physical Activity
Description: Physical activity is determined using daily mean amplitude deviation in milligrams by wrist worn accelerometer over a period of approximately 7 days within late pregnancy (35-37 weeks gestation). Mean amplitude deviation describes the mean distance of data points from the mean, and higher values denote higher levels of physical activity.
Time Frame: Approximately 7 days within 35-37 weeks gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 36 | 8 | 10 | 0
milligrams | 47.5 (11.4) | 52.9 (10.7) | 41.4 (12.6) |

4. Secondary Outcome: Energy Expenditure During Sleep
Description: Energy expenditure during sleep is determined by 1 overnight stay in a whole body calorimeter within early pregnancy (13-16 weeks gestation).
Time Frame: 1 day within 13-16 weeks gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 36 | 8 | 10 | 0
kilocalories per day | 1648 (198) | 1688 (218) | 1907 (329) |

5. Secondary Outcome: Energy Expenditure During Sleep
Description: Energy expenditure during sleep is determined by 1 overnight stay in a whole body calorimeter within late pregnancy (35-37 weeks gestation).
Time Frame: 1 day within 35-37 weeks gestation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 36 | 8 | 10 | 0
kilocalories per day | 1975 (216) | 2081 (288) | 2125 (278) |

6. Secondary Outcome: Percentage of Protein of Energy Intake
Description: Percentage of protein of energy intake is determined by remote food photography method within early pregnancy (13-16 weeks gestation).
Time Frame: Approximately 7 days within 13-16 weeks gestation
Population: Analysis could not be completed for the Arm (Pregnant Women Not Included in Analysis) for various reasons. In the analyzed Arms, some participants were not analyzed as energy intake by remote food photography method was less than 60% of the total energy expenditure during that period.
Measure: Mean (Standard Deviation); unit: percentage of energy intake
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 29 | 5 | 5 | 0
percentage of energy intake | 15.3 (3.8) | 16.3 (3.6) | 18.9 (12.1) |

7. Secondary Outcome: Percentage of Protein of Energy Intake
Description: Percentage of protein of energy intake is determined by remote food photography method within late pregnancy (35-37 weeks gestation).
Time Frame: Approximately 7 days within 35-37 weeks gestation
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of energy intake
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 29 | 5 | 5 | 0
percentage of energy intake | 15.3 (4.3) | 16.1 (3.8) | 13.7 (3.1) |

8. Secondary Outcome: Percentage of Fat of Energy Intake
Description: Percentage of fat of energy intake is determined by remote food photography method within early pregnancy (13-16 weeks gestation).
Time Frame: Approximately 7 days within 13-16 weeks gestation
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of energy intake
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 29 | 5 | 5 | 0
percentage of energy intake | 38.1 (4.3) | 38.0 (5.8) | 34.0 (5.6) |

9. Secondary Outcome: Percentage of Fat of Energy Intake
Description: Percentage of fat of energy intake is determined by remote food photography method within late pregnancy (35-37 weeks gestation).
Time Frame: Approximately 7 days within 35-37 weeks gestation
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of energy intake
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 29 | 5 | 5 | 0
percentage of energy intake | 38.3 (5.9) | 39.6 (6.0) | 34.6 (5.6) |

10. Secondary Outcome: Percentage of Carbohydrate of Energy Intake
Description: Percentage of carbohydrate of energy intake is determined by remote food photography method within early pregnancy (13-16 weeks gestation).
Time Frame: Approximately 7 days within 13-16 weeks gestation
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of energy intake
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 29 | 5 | 5 | 0
percentage of energy intake | 47.6 (7.0) | 46.6 (8.5) | 48.2 (12.3) |

11. Secondary Outcome: Percentage of Carbohydrate of Energy Intake
Description: Percentage of carbohydrate of energy intake is determined by remote food photography method within late pregnancy (35-37 weeks gestation).
Time Frame: Approximately 7 days within 35-37 weeks gestation
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of energy intake
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
Number analyzed (Participants) | 29 | 5 | 5 | 0
percentage of energy intake | 47.4 (8.6) | 44.9 (8.0) | 52.7 (8.3) |

ADVERSE EVENTS:
Time Frame: 1 year 6 months
Arm/Group | Pregnant Women With Excess Gestational Weight Gain | Pregnant Women With Recommended Gestational Weight Gain | Pregnant Women With Inadequate Gestational Weight Gain | Pregnant Women Not Included in Analysis
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/8 | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 3/36 | 1/8 | 0/10 | 4/18
Other Adverse Events (participants affected / at risk) | 36/36 | 7/8 | 9/10 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnant Women With Excess Gestational Weight Gain (N=36) | Pregnant Women With Recommended Gestational Weight Gain (N=8) | Pregnant Women With Inadequate Gestational Weight Gain (N=10) | Pregnant Women Not Included in Analysis (N=18)
Miscarriage or Pregnancy Loss (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hip pain requiring surgery
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Aphasia requiring overnight hospital stay
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Kidney infection requiring hospital stay of 3 nights.
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Vertigo requiring hospital stay.
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pelvic infection which caused preterm premature rupture of membranes and required a hospital stay.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnant Women With Excess Gestational Weight Gain (N=36) | Pregnant Women With Recommended Gestational Weight Gain (N=8) | Pregnant Women With Inadequate Gestational Weight Gain (N=10) | Pregnant Women Not Included in Analysis (N=18)
Cold/sinus congestion (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 2 (3) | 4 (5) | 3 (3)
Headaches (Nervous system disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Heartburn (Gastrointestinal disorders) | 7 (8) | 1 (1) | 4 (4) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 4 (4) | 2 (2) | 1 (1)
Gestational Diabetes (Endocrine disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 7 (8) | 2 (2) | 5 (5) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Allergies (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Fungal Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacterial Infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Body Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Stomach virus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fainting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal Tunnel (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folate Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cystic Hygroma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Eighteen women who enrolled in the study were not included in analysis for various reasons. The reasons included: missing data from 13-16 gestational week visit, miscarriage, lost to follow-up, preterm delivery, pre-eclampsia, unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT01954342/Prot_SAP_000.pdf